CLINICAL TRIAL: NCT04880577
Title: Tenofovir Alafenamide for Treatment of Symptoms and Neuroprotection in Relapsing Remitting Multiple Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Michael, Levy M.D.,Ph.D., Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P003311
Record Dates: First submitted 2021-04-30; First posted 2021-05-10 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Fatigue
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Fatigue | interventions — Tablets; tenofovir alafenamide; ocrelizumab; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAF (Experimental): 25 mg of daily TAF
  Interventions: Drug: TENOFOVIR ALAFENAMIDE FUMARATE 25 Mg ORAL TABLET [VEMLIDY]
- Placebo (Placebo Comparator): Placebo pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TENOFOVIR ALAFENAMIDE FUMARATE 25 Mg ORAL TABLET [VEMLIDY] — The study is designed to add on TAF to anti-CD20 therapies
  Other Names: Ocrelizumab; rituximab
  Arms: TAF
Drug: Placebo — Placebo arm
  Other Names: ocrelizumab; rituximab
  Arms: Placebo

SUMMARY:
As the in vivo reservoir of the Epstein-Barr virus, B cells play an important role in the perpetuation of MS disease activity. B cell depletion therapy with medications like ocrelizumab or rituximab have proved very successful in preventing clinical relapses and MRI activity in MS, but incomplete in terms of neuroprotection and symptomatic outcomes. Ocrelizumab and rituximab only target naïve and memory B cells expressing the CD20 marker but do not deplete the wide spectrum of B cell lineages including plasmablasts and plasma cells, which are also key reservoirs for EBV. This is particularly relevant to the mechanism of action of TAF, since EBV lytic reactivation occurs in coordination with B-cell differentiation. In vivo, the initiation of plasma cell differentiation provides the physiological trigger for EBV lytic reactivation, and EBV utilizes the plasma cell differentiation program to replicate. As these cells are ineffectively depleted by anti-CD20 treatment, the use of TAF would be highly complementary as an add-on treatment to anti-CD20 therapy.

Anti-EBV therapy with TAF in combination with ocrelizumab or rituximab will therefore provide a synergistic approach to cover the whole EBV reservoir.

The primary aims of the proposed trial are to determine if TAF, at the standard dose of 25 mg/day administered for 12 months:

i) is safe and well-tolerated by individuals with RRMS over a period of treatment of 12 months; ii) leads to an overall improvement in fatigue, as assessed by the Modified Fatigue Impact Scale by 12 months; and iii) causes a reduction in serum concentrations of neurofilament light chain (NfL), a marker of neuronal damage in MS.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness and ability to comply with all study procedures and availability for the duration of the study
3. Aged 18+ years
4. Diagnosis of MS using revised 2010 McDonald criteria of clinically definite MS.
5. Receiving treatment with either ocrelizumab or rituximab on a regular twice-yearly schedule. The first infusion must have been received at least 6 months before enrollment.
6. Must report significant fatigue during the past 3 months not due to a cause other than MS.
7. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.
8. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.

Exclusion Criteria:

1. Pregnancy or lactation
2. Known allergic reactions to components of TAF
3. Treatment with another investigational drug or other MS-directed intervention such as glatiramer acetate, or dimethyl fumarate within 3 months
4. Positive HIV antibody test, active or latent hepatitis B
5. Relapse and/or steroid treatment within the previous 30 days
6. Baseline EDSS > 7
7. Current symptoms of severe, progressive, or uncontrolled renal, hematologic, gastrointestinal, pulmonary, cardiac, or neurologic disease, or other medical conditions that, in the opinion of the Investigator, might place the subject at unacceptable risk for participation in this study
8. Known history of sleep apnea, narcolepsy, or other significant sleep disorders
9. Recent changes to medications affecting sleep or fatigue or changes in dosage of those medications within 90 days
10. Creatinine clearance (CrCl) <55mL/min, as calculated by the Cockcroft-Gault equation
11. Taking medication with known interactions with tenofovir alafenamide including: Acyclovir, valacyclovir, adefovir, cabozantinib, carbamazepine, cidofovir, cladribine, cobicistat, diclofenac, multiple NSAIDs or chronic high dose NSAIDs, fosphenytoin or phenytoin, ganciclovir, valganciclovir, oxcarbazepine, phenobarbital, primidone, rifabutin, rifampin, rifapentine, sofosbuvir, tipranavir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2024-02-14 (Estimated); Study Completion 2025-02-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From baseline to 12 months
  Safety and tolerability of TAF by individuals with RRMS
Modified Fatigue Impact Scale | From baseline to 12 months
  Change in Modified Fatigue Impact Scale (MFIS) score (range 0-84, higher is more fatigue)
serum concentrations of neurofilament light chains (NfL) | From baseline to 12 months
  Reduction in serum concentrations of neurofilament light chains (NfL), a marker of neuronal damage in MS (pg/ml, the higher the more neuronal damage)

SECONDARY OUTCOMES:
Multiple Sclerosis Impact Scale-29 | From baseline to 12 months
  Change in Multiple Sclerosis Impact Scale-29 (MSIS-29) score (range 0-100, higher scores are more impactful)
Short Form 36 Health Survey Questionnaire | From baseline to 12 months
  Change in Short Form 36 (SF-36) Health Survey Questionnaire (range 0-100, higher scores are healthier)
Beck Depression Inventory | From baseline to 12 months
  Change in Beck Depression Inventory (BDI-II) score (range 0-63, higher score indicate more severe depression)
Perceived Deficits Questionnaire | From baseline to 12 months
  Change in Self-Reported Cognitive Dysfunction: Perceived Deficits Questionnaire (PDQ)(range 0-80, higher scores indicate more perceived cognitive dysfunction)
Annualized relapse rate | From baseline to 12 months
  Number of relapses per year
Expanded Disability Status Scale | From baseline to 12 months
  Change in Expanded Disability Status Scale (EDSS) score (range 0-10, higher scores are more disabled)
Symbol Digit Modality Test | From baseline to 12 months
  Change in Symbol Digit Modality Test (SDMT)
Timed 25 Foot Walk | From baseline to 12 months
  Change in Timed 25 Foot Walk Test (T25-FW) (timed in seconds, longer time is more disabled)
9-Hole Peg Test | From baseline to 12 months
  Change in 9-Hole Peg Test (9-HPT)
Number of new MRI lesions | From baseline to 12 months
  New active MRI lesions (gadolinium-enhancing, and new or enlarging T2 lesions)
EBV viral load | From baseline to 12 months
  Change in EBV viral load in saliva
EBV titers | Comparison of baseline to 6 months and 12 months
  Change in anti-EBV antibody titers

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levy, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No